CLINICAL TRIAL: NCT05843747
Title: Ex Vivo Transformation of White Adipose Tissue (WAT) Into Brown Adipose Tissue (BAT) in Morbidly Obese Patients Using the Ex Vivo Adipocyte Expansion (ExAdEx) Approach: Proof of Concept. From White to Brown Adipose Tissue
Acronym: OBADEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-AOIP-04
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sampling (Experimental)
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — During thier bariatric surgery, samples of adipose tissue will be done

SUMMARY:
Obesity and metabolic associated diseases such as type 2 diabetes, NASH, cardiovascular diseases, are the dysregulation of energy homeostasis associated with an imbalance between different types of adipose tissues (ATs). White AT (WAT) which stores energy and functions as a fat storage depot, is fibrotic whith chronic inflammation and is found in excess. On the other hand, brown and beige ATs (BATs), considered as the good ATs because they regulate energy expenditure, are almost undetectable in individuals with obesity. In addition, BAT and WAT produce different hormones that are involved in the control of energy homeostasis via central and peripheral actions. A promising emerging therapeutic approach is to restore BAT in patients with severe obesity in two ways, i) by stimulating BAT in individuals with obesity by pharmacological treatment, ii) by injecting BAT into individuals with obesity using a cell-based therapy approach. However, the development of these two proposals is limited both by the lack of in vitro preclinical BAT models relevant for the screening and validation stages of drug candidates, and by the lack of physiologically functional BAT compatible with tissue graft. The bottleneck is the absence of an unlimited source of human BAT.

The ExAdEX technology makes possible in vitro to turn WAT derived from lean donors into BAT. This new technology offers the possibility of having in vitro predictive human 3D models suitable for the identification and characterization of compounds affecting AT biology, and paves the way for the production of BAT for cell-based therapy of obesity and associated metabolic diseases.

The Primary objective of the study is addressed the effectiveness of the ExAdEx process to induce, ex vivo, the conversion of WAT from obese patients into TAB. The secondary objectives are 1) to compare the efficacy for conversion into BAT when WAT derived from either from visceral or from subcutaneous AT; 2) to investigate the capacity of the ExAdEX-BAT to produce the FGF21 and adiponectin batokines and to respond to insulin.

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

* Karnofsky index > 70
* IMC > 35 kg/m2 associated with a comorbidity : hypertension ; type 2 diabetes; disabling osteoarthritis; sleep apnea syndrome with device.
* Failure of a previous well-conducted medical treatment (multidisciplinary management of more than six months preoperatively)

Exclusion Criteria:

* Psychiatric counter-indications
* Anaesthetic counter-indications
* Progressive neoplastic pathologies
* Chronic alcoholism
* Severe uncontrolled infection
* Renal failure (Cockroft's clearance <30ml/min)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
WAT/TAB conversion | At 1 month
  WAT/BAT conversion efficiency based on the expression level of the UCP1 marker in the cultures

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Archet 2, Nice, Alpes-Mritimes, France

IPD SHARING:
Plan to Share IPD: No